CLINICAL TRIAL: NCT03533660
Title: Alcohol Biosensor Monitoring for Alcoholic Liver Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Andrea DiMartini, Professor of Psychiatry and Surgery, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R21AA025730 (NIH); R21AA025730 (NIH)
Record Dates: First submitted 2018-04-13; First posted 2018-05-23 (Actual); Results first posted 2022-11-07 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Alcohol Use, Unspecified
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Intervention Model Description: RCT feedback vs. enhanced usual care
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Feedback (Active Comparator): Participant will receive a brief feedback on data downloaded from the ABM and information about treatment resources
  Interventions: Behavioral: Feedback
- Enhanced usual care (Active Comparator): Participant will receive information about remaining abstinent and about treatment resources
  Interventions: Behavioral: Enhanced Usual Care

INTERVENTIONS:
Behavioral: Feedback — Participant will receive a brief feedback on alcohol use data downloaded from the ABM and information about treatment resources
  Arms: Feedback
Behavioral: Enhanced Usual Care — Participant will receive information on self reported alcohol use and information about remaining abstinent and about treatment resources
  Arms: Enhanced usual care

SUMMARY:
Successful treatment of alcohol associated liver disease (AALD) depends primarily on abstinence from alcohol. The investigators propose a randomized clinical trial of alcohol biosensor monitoring for patients with alcohol associated liver disease to determine if monitoring with feedback on alcohol use patterns reduces alcohol consumption and improves outcomes.

DETAILED DESCRIPTION:
The investigators propose a 3 month randomized controlled trial (RCT) pilot of alcohol biosensor monitoring (ABM)(WrisTAS) for patients with Alcohol Associated Liver Disease (AALD) who intend to stop drinking. All participants will wear the ABM device but participants will be randomized to receive either personalized feedback on the data recorded on the device (n=30) or enhanced usual care without feedback on device data (n=30). The investigators will determine whether ABM plus feedback improves outcomes for AALD patients compared to enhanced usual care and hypothesize ABM feedback will reduce alcohol consumption, improve motivation and self-efficacy for abstinence and improve engagement in treatment. The investigators will also conduct research including qualitative data collected from participants who will provide opinions on ABM feasibility, acceptability, and usability. Qualitative methods are especially useful for understanding the perceived needs, barriers, and preferences for monitoring alcohol use and are especially required for future translation of this technology into clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients with AALD followed at our liver disease clinic,
* 18 years or older,
* willing to accept randomization,
* and agree to wear device for 3 months,
* SOCRATES problem recognition subscale score >26 (scores <26 indicate very low recognition of an alcohol problem).

Exclusion Criteria:

* Non-English speaking,
* Montreal Cognitive Assessment (MOCA) scores <21 (moderate cognitive impairment) or neurologic diseases (e.g. Parkinson's),
* patients with unresponsive acute alcoholic hepatitis, multi-organ failure, fulminant hepatic failure,
* cancer/terminal illness;
* those unable to wear a wrist monitor (e.g., edema);
* lacking a residence, or unable to identify a contact person (if lost to follow-up).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2018-09-13 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea DiMartini, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
The study database will be reviewed to ensure that no identifying information of any type is contained therein. A downloadable, de-identified data set and data dictionary will be made available electronically from the PI after the request is reviewed by the research team for scientific merit and requestors provide evidence to the PI that (a) their plan for the use of such data has been approved by their institution's Institutional Review Board or its equivalent, and (b) they have completed NIH requirements for training in research integrity and human subjects protection.
Time Frame: To provide the investigators adequate time to prepare and submit the majority of publications likely to result from the research, data obtained from the study will be made publicly available no sooner than 18 months after the conclusion of the study.
Access Criteria: Access can be requested from PI following plan description and time frame noted above

REFERENCES:
- [Derived] DiMartini A, Behari J, Dunn M, Bataller RA, Jakicic JM, McNulty M, Young RC, Dew MA. Challenges and Solutions for Monitoring Alcohol Use in Patients With Alcohol-Related Liver Disease: Pilot Study of a Wearable Alcohol Biosensor. Psychosom Med. 2023 Sep 1;85(7):596-604. doi: 10.1097/PSY.0000000000001203. Epub 2023 Apr 17. PMID 37097109

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Feedback | Enhanced Usual Care
Started | 15 | 18
Completed | 11 | 10
Not Completed | 4 | 8
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Death | 2 | 4
Not completed — Adverse Event | 0 | 2

BASELINE CHARACTERISTICS:
Population: These 27 participants are those that went through the initial intake assessment and thus are included in the analyses
Groups:
- Total: Total of all reporting groups
Arm/Group | Feedback | Enhanced Usual Care | Total
Number analyzed (Participants) | 14 | 13 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 43 (10) | 47 (10) | 45 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 16
  Male | 5 | 6 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 14 | 12 | 26
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 14 | 11 | 25
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Alcohol Use
Description: Average number of drinks per drinking episode per interval (month) of device wear. We analyzed the number of drinks per drinking episode and present the group average per month interval of assessment.
Time Frame: continuous for up to 3 months
Population: We analyzed data for all 27 participants. Only 6 participants drank alcohol and their data is shown below. The remaining 21 participants had no alcohol use data to present.
Measure: Mean (Standard Deviation); unit: drinks per episode
Groups:
- Feedback: These data are only on those in the feedback group who drank
- Enhanced Usual Care: These data are only on those in the EUC group who drank
Arm/Group | Feedback | Enhanced Usual Care
Number analyzed (Participants) | 0 | 6
drinks per episode
  Average drinks per drinking episode for first interval (month) of device wear |  | 7.4 (3.7)
  Average drinks per drinking episode for second interval (one month) of device wear: number analyzed (Participants) | 0 | 4
  Average drinks per drinking episode for second interval (one month) of device wear |  | 5.3 (3.9)
  Average drinks per drinking episode for third interval (one month) of device wear: number analyzed (Participants) | 0 | 4
  Average drinks per drinking episode for third interval (one month) of device wear |  | 4.4 (3.5)

2. Primary Outcome: Percent of Days Drinking Per Interval of Device Wear
Description: Percent of days drinking per interval of device wear: We analyzed the data by number of drinking episodes per individual per days of device wear and present the mean percent days drinking per assessment interval
Time Frame: 3 months
Population: We analyzed all 27 participants but only 6 participants were found to be drinking. Thus only participants who drank (n=6) were analyzed for drinking outcomes. The numbers at follow up assessments are different than initially enrolled due to drop out
Measure: Mean (Standard Deviation); unit: percentage of days drinking
Groups:
- Feedback: These data relate to only those in the Feedback group who drank
- Enhanced Usual Care: These data relate to only those in the EUC group who drank
Arm/Group | Feedback | Enhanced Usual Care
Number analyzed (Participants) | 0 | 6
percentage of days drinking
  % Days of drinking per first interval of device wear |  | 0.48 (0.48)
  % Days of drinking per second interval of device wear: number analyzed (Participants) | 0 | 4
  % Days of drinking per second interval of device wear |  | 0.74 (0.16)
  % Days of drinking per third interval of device wear: number analyzed (Participants) | 0 | 4
  % Days of drinking per third interval of device wear |  | 0.42 (0.34)

3. Secondary Outcome: Improved Readiness for Alcohol Abstinence and Initiation of Change
Description: Stages of Change Readiness & Treatment Eagerness Scale (SOCRATES) is a 19-item instrument that measures readiness for change assessing three areas; ambivalence, recognition, and taking steps with change scores assessing the impact of an intervention on these areas. Three subscale scores are produced with total scores ranging 19-95 and higher score indicating greater readiness:
  * 7 items for recognition of an alcohol problem (scores range from low of 7 to highest of 35)
  * 4 items for ambivalence (range from low of 4 to highest of 20)
  * 8 items for taking steps to make a positive change in drinking (range from low of 8 to highest of 40)
Time Frame: Scores determined at initiation, 6 weeks and 3 months of participation
Population: numbers at follow up assessments are different than initially enrolled due to drop out
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Feedback | Enhanced Usual Care
Number analyzed (Participants) | 14 | 13
score on a scale
  SOCRATES Total Score: Intake assessment | 82 (7) | 79 (14)
  Subscale Recognition: intake | 32 (3) | 31 (6)
  Subscale Ambivalence: intake | 14 (5) | 13 (4)
  Subscale Taking Steps: intake | 35 (3) | 34 (5)
  SOCRATES Total Score: 6 week assessment: number analyzed (Participants) | 12 | 11
  SOCRATES Total Score: 6 week assessment | 72 (9) | 77 (13)
  Subscale Recognition: 6 weeks: number analyzed (Participants) | 12 | 11
  Subscale Recognition: 6 weeks | 27 (5) | 31 (6)
  Subscale Ambivalence: 6 weeks: number analyzed (Participants) | 12 | 11
  Subscale Ambivalence: 6 weeks | 9 (4) | 13 (4)
  Subscale Taking Steps: 6 weeks: number analyzed (Participants) | 12 | 11
  Subscale Taking Steps: 6 weeks | 28 (5) | 33 (4)
  SOCRATES Total Score: 3 Month assessment: number analyzed (Participants) | 11 | 10
  SOCRATES Total Score: 3 Month assessment | 70 (6) | 73 (15)
  Subscale Recognition: 3 months: number analyzed (Participants) | 11 | 10
  Subscale Recognition: 3 months | 24 (5) | 28 (7)
  Subscale Ambivalence: 3 months: number analyzed (Participants) | 11 | 10
  Subscale Ambivalence: 3 months | 9 (4) | 13 (5)
  Subscale Taking Steps: 3 months: number analyzed (Participants) | 11 | 10
  Subscale Taking Steps: 3 months | 28 (4) | 31 (5)
Statistical Analysis 1: Comparison: Feedback vs Enhanced Usual Care; Test type: Superiority; p < .05, t-test, 2 sided — Applies to SOCRATES subscales recognition, ambivalence, taking steps at 6 weeks
Statistical Analysis 2: Comparison: Feedback vs Enhanced Usual Care; Test type: Superiority; p > .05, t-test, 2 sided — Applies to SOCRATES total scores and subscales (recognition, ambivalence, and taking steps) at intake and 3 months

4. Secondary Outcome: Self Efficacy to Remain Abstinent
Description: Alcohol Abstinence Self-efficacy (AASE) evaluates confidence in ability to abstain from drinking in situations that represent typical drinking cues. Four subscales with 5 specific situations each are rated on confidence not to drink in each situations on a 5-point Likert scale from 1=not at all confident to 5=extremely confident. Total scores range from 20-100 with higher scores reflecting greater self confidence not to drink.
  * negative affect situations (range from low confidence of 5 to highest confidence of 25)
  * social/positive situations (range from low confidence of 5 to highest confidence of 25)
  * physical and other concerns situations (range from low confidence of 5 to highest confidence of 25)
  * cravings and urges situations (range from low confidence of 5 to highest confidence of 25)
Time Frame: Scores determined at initiation, 6 weeks and 3 months of participation
Population: numbers at follow up assessments are different than initially enrolled due to drop out
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Feedback | Enhanced Usual Care
Number analyzed (Participants) | 14 | 13
score on a scale
  Alcohol Self Efficacy Scale: Intake assessment | 82 (15) | 85 (25)
  Subscale Negative Affect: intake | 20 (5) | 21 (7)
  Subscale Social Positive: intake | 21 (4) | 21 (7)
  Subscale Physical Concern: intake | 22 (3) | 22 (6)
  Subscale Withdrawal Urges: intake | 19 (5) | 22 (6)
  Alcohol Self Efficacy Scale: 6 week assessment: number analyzed (Participants) | 12 | 11
  Alcohol Self Efficacy Scale: 6 week assessment | 88 (10) | 83 (26)
  Subscale Negative Affect: 6 weeks: number analyzed (Participants) | 12 | 11
  Subscale Negative Affect: 6 weeks | 21 (3) | 20 (7)
  Subscale Social Positive: 6 weeks: number analyzed (Participants) | 12 | 11
  Subscale Social Positive: 6 weeks | 23 (3) | 20 (7)
  Subscale Physical Concern: 6 weeks: number analyzed (Participants) | 12 | 11
  Subscale Physical Concern: 6 weeks | 23 (2) | 21 (6)
  Subscale Withdrawal Urges: 6 weeks: number analyzed (Participants) | 12 | 11
  Subscale Withdrawal Urges: 6 weeks | 21 (3) | 21 (6)
  Alcohol Self Efficacy Scale: 3 month assessment: number analyzed (Participants) | 11 | 10
  Alcohol Self Efficacy Scale: 3 month assessment | 91 (11) | 77 (30)
  Subscale Negative Affect: 3 months: number analyzed (Participants) | 11 | 10
  Subscale Negative Affect: 3 months | 22 (4) | 20 (7)
  Subscale Social Positive: 3 months: number analyzed (Participants) | 11 | 10
  Subscale Social Positive: 3 months | 23 (3) | 18 (9)
  Subscale Physical Concern: 3 months: number analyzed (Participants) | 11 | 10
  Subscale Physical Concern: 3 months | 24 (2) | 20 (6)
  Subscale Withdrawal Urges: 3 months: number analyzed (Participants) | 11 | 10
  Subscale Withdrawal Urges: 3 months | 23 (3) | 19 (8)
Statistical Analysis 1: Comparison: Feedback vs Enhanced Usual Care; Test type: Superiority; p > .05, t-test, 2 sided — Applies to alcohol self-efficacy scale total score and subscales scores at intake, 6 weeks and 3 months

5. Secondary Outcome: Medical Outcomes
Description: AALD related hospitalizations and ER visits - total count of participants in each arm who experienced these outcomes
Time Frame: Counts determined at initiation, 6 weeks and 3 months of participation
Population: Two participants in the EUC arm had died by the 3 month assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Feedback | Enhanced Usual Care
Number analyzed (Participants) | 14 | 13
Participants
  Intake assessment: Count of participants hospitalized in prior 90 days | 14 | 12
  Intake assessment: Count of participants in emergency room in prior 90 days | 5 | 2
  6 week assessment: Count of participants hospitalized between intake and 6 week assessment | 6 | 6
  6 week assessment: Count of participants in emergency room between intake and 6 week assessment | 4 | 5
  3 month assessment: Count of participants hospitalized between 6 week and 3 month assessment: number analyzed (Participants) | 14 | 11
  3 month assessment: Count of participants hospitalized between 6 week and 3 month assessment | 2 | 2
  3 month assessment: Count of participants in emergency room between 6 week and 3 month assessment: number analyzed (Participants) | 14 | 11
  3 month assessment: Count of participants in emergency room between 6 week and 3 month assessment | 2 | 3

6. Secondary Outcome: Qualitative Interviews
Description: Qualitative interviews of participants will use a semi-structured script of open-ended stem questions with prompts. The qualitative assessment will cover such topics as patients' perceived need/psychologic barriers (e.g., beliefs in value of ABM in their clinical care and for their relationship with clinicians) and experience with ABM (e.g., wearability, satisfaction, and barriers to monitoring). Transcribed interviews will be thematically coded. The constant comparison method will be used, and subsequent interviews may be modified/informed by findings from previous interviews to explore emerging themes as the analysis proceeds.
Time Frame: measured at three months (completion of the participants use of ABM)
Population: Includes 21 participants who completed the study and 2 additional participants who had to withdraw prior to completing the full study but were able to complete the qualitative interview. The purpose of qualitative interviews was to determine themes across both groups not between groups. We assigned qualitative data its own separate purpose within the larger project. We did not plan to quantitatively analyze the qualitative data.
Measure: Number; unit: Themes
Groups:
- All Participants: Positive and negative themes that emerged from qualitative data analyses on usability, acceptability, feasibility, efficiency, impact of device on behaviors, preference or barriers from interviews with all participants
Arm/Group | All Participants
Number analyzed (Participants) | 23
Themes
  Positive Usability examples: comfortable, no interference activities/lifestyle/sleep, easy to wear | 6
  Positive Acceptability example: looks didn't bother, didn't feel self-conscious, didn't hide purpose | 8
  Positive Feasibility examples: willing to wear, didn't take off, wouldn't change dr relationship | 7
  Positive Efficiency examples: benefit if prescribed, improve honesty, more data/ better/ accurate | 6
  Positive Impact of device on behavior examples: visual deterrent, accountability, therapeutic value | 10
  Positive Preferences, Facilitators, or Barriers: helpful if dr prescribed, gives proof not drinking | 9
  Negative Usability examples: uncomfortable/cumbersome/annoying, interfered with sleep | 7
  Negative Acceptability examples: conspicuous, felt self-conscious, appearance not optimal | 4
  Negative Feasibility examples: had to take off for a lot of activities/ to avoid damaging | 6
  Negative Efficiency examples: Wouldn't improve medical care, already honest about alcohol use | 2
  Negative Impact of device on behavior examples: can't prevent drinking, have to buy into concept | 5
  Negative Preferences, Facilitators, or Barriers: potential negative feelings/stigma/reminder | 8

ADVERSE EVENTS:
Time Frame: Data was collected over the three month period that the participants participated in the study.
Description: We collected data only on those who completed the intake interview and participated in the study (n=27). Data was collected from medical record review and information on device wearing issues was collected during monthly assessments. We tracked mortality, and number of hospitalizations and emergency room visits but our protocol was not to identify the causes/reasons for ER visit/hospitalizations. There were no serious adverse events related to the study.
Arm/Group | Feedback | Enhanced Usual Care
All-Cause Mortality (participants affected / at risk) | 2/14 | 2/13
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/13
Other Adverse Events (participants affected / at risk) | 7/14 | 7/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Feedback (N=14) | Enhanced Usual Care (N=13)
skin irritation/indentation (Skin and subcutaneous tissue disorders) | 7 (7) | 7 (7) — Number of participants who reported skin irritation/indentation typically noted this was from wearing the device too tightly - strap was adjustable and most reported issues resolved with adjustment/removal
strap being itchy/scratchy (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (4) — Number of participants who reported device strap was itchy/scratchy
Uncomfortable (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2) — Number of participants who reported wearing the device was uncomfortable (sleeping or otherwise)
Participants uncomfortable with device appearance (Product Issues) | 1 (1) | 2 (2) — Number of participants who commented that the device was unappealing in appearance

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-15): https://cdn.clinicaltrials.gov/large-docs/60/NCT03533660/Prot_SAP_000.pdf